CLINICAL TRIAL: NCT01567800
Title: A Feasibility Study of Hypoxia Imaging in Patients With Prostate Cancer Using Positron Emission Tomography (PET) With 18F-Fluoroazomycin Arabinoside (18F-FAZA)
Brief Title: Prostate Hypoxia FAZA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: UHN REB 11-0953-C
Record Dates: First submitted 2012-03-23; First posted 2012-03-30 (Estimated); Last update posted 2025-02-10 (Actual); Status verified 2025-02

CONDITIONS: Prostate Cancer
Keywords: Procedure/Surgery: 18F-Fluoroazomycin Arabinoside (18F-FAZA)
MeSH Terms: conditions — Prostatic Neoplasms | interventions — fluoroazomycin arabinoside

ARMS (1):
- PET FAZA imaging (Experimental): PET FAZA imaging of tumor hypoxia in patients with prostate cancer
  Interventions: Other: 18F-Fluoroazomycin Arabinoside (18F-FAZA)

INTERVENTIONS:
Other: 18F-Fluoroazomycin Arabinoside (18F-FAZA) — PET scan with the radiolabelled tracer 18F-FAZA

SUMMARY:
The purpose of this study is to look for low levels of oxygen (hypoxia) in prostate cancer using a special x-ray test called a positron emission tomography (PET)scan. Hypoxia may have an effect on how prostate cancer grows and responds to treatments like radiotherapy and chemotherapy. The use of PET scans to measure hypoxia may be better and simpler than the methods used previously.

ELIGIBILITY:
Inclusion Criteria:

* Age => 18 years
* Histologic diagnosis of adenocarcinoma of the prostate
* Bulky intermediate risk, high risk or metastatic prostate cancer

Bulky intermediate risk: cT1-2 with >50% of diagnostic biopsy cores containing cancer and Gleason 6 or 7 and prostate specific antigen (PSA) >10 and ≤20 OR

High risk:

cT1-2 with Gleason score ≥8; or cT1-2 with PSA >20; or cT3 OR N+ and/or M1 disease OR Newly diagnosed hormone-refractory prostate cancer - Intention to treat using radiotherapy +/- concurrent and adjuvant hormonal therapy

* Intention to treat with radiotherapy, hormonal therapy, other systemic treatment for prostate cancer, or a combination of these according to the Princess Margaret Genitourinary Site policies.
* Previous or concurrent anti-cancer therapy for the PET FAZA target lesion allowed
* Ability to provide written informed consent to participate in the study

Exclusion Criteria:

* Inability to lie supine for more than 60 minutes
* Patients taking the drug disulfiram (Antabuse)
* Contraindications for MRI: only applicable in cases where the PET FAZA target lesion is identified as the prostate gland. Patients with target lesions at other anatomic sites will not undergo MR imaging.
* Patients weighing > 136 kg

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2012-04; Primary Completion 2027-06 (Estimated); Study Completion 2028-03 (Estimated)

PRIMARY OUTCOMES:
Number of patients treated with the PET tracer FAZA to image primary tumor hypoxia in patients with prostate cancer prior to treatment with radiotherapy +/- concurrent and adjuvant hormonal therapy | 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- University Health Network, Toronto, Ontario, Canada